CLINICAL TRIAL: NCT05870826
Title: Pilot Study on the Effects of MLS (Multiwave Locked System) LASER Therapy in Patients With Chronic Nonspecific Low Back Pain: Randomized Controlled Trial Versus Placebo
Brief Title: The Effects of MLS LASER Therapy in Patients With Chronic Nonspecific Low Back Pain
Acronym: MLSLASERlumb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Mariagrazia Benedetti, Head of the Unit of Physical Medicine and Rehabilitation, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0012596
Record Dates: First submitted 2022-06-27; First posted 2023-05-23 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Non-specific Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham laser therapy (Sham Comparator): The control group (PL group) is subjected to a laser sham (placebo), employing a device identical to the one under investigation but lacking the laser emission capability, and the same mode of administration in terms of time and place. Both the sham laser and the test device emit visible light of the same color and are not distinguishable in any way.
  Interventions: Other: Sham laser therapy
- Laser therapy (Experimental): The MLS group receives MLS synchronized diode laser therapy emitted by the MLS M8 robotic device (ASA, Italy).
  MLS M8 (ASA, Arcugnano, Italy), a Class IV (high-power) laser approved by the Food Drug Administration (FDA) and CE certified, characterized by a combined, synchronized two-wavelength (CPW) emission: a continuous emission with a wavelength of 808 nm and a pulsed emission at 905 nm.
  The duration of each session is 5 min 45 sec.seconds, delivering a total energy of 1500 J and an energy dose of 5 J/cm2, for an area of 300 cm2.
  The robotic device is placed in the lumbar area, oriented on the muscles erector spinae and quadratus lumborum. The target area set on the device is "lumbar area." The parameters set on the device are "Synchronized Emission of Continuous Pulsed Wave (CPW)," "intensity of 100%," "time of 5 minutes and 45 seconds," and "area of 1x300 cm2."
  Interventions: Other: Multiwave locked system laser therapy

INTERVENTIONS:
Other: Multiwave locked system laser therapy — High intensity laser therapy
  Arms: Laser therapy
Other: Sham laser therapy — Sham laser therapy
  Arms: Sham laser therapy

SUMMARY:
Non-specific cronic low back pain is very common condition affecting 80-85% of adults. The most common therapies for low back pain are: patient education, excercise and physical therapy. High intensity laser therapy has been shown to be an effective treatment to improve sympthoms in patient with non-specific low back pain when combined wth exercise.

The aim of this study is to assess the effects of a multi-wave locked system laser therapy in patient with non-specif low back pain when administered alone.

DETAILED DESCRIPTION:
Chronic nonspecific low back pain, given its high prevalence globally and the disability resulting from it, results in significant deterioration in quality of life and substantial both social and economic costs. The determinants are predominantly biological, in particular musculoskeletal alterations of the lumbar region, but psychosocial factors also contribute significantly to the manifestation of the disorder.

Patients with chronic nonspecific low back pain are characterized by pain intensity sometimes disabling, a reduction in lumbar range of motion (ROM) and the frequent absence of flexion-relaxation phenomenon (FRP). Both high-power and low-power laser therapy, especially when included in a multidimensional rehabilitation plan, seems effective in improving both pain and function of affected patients. MLS (Multiwave Locked System) laser therapy is an innovative high-power technology characterized by the combined and synchronized emission of laser light at two wavelengths (a continuous emission with a wavelength wavelength of 808 nm and a pulsed emission at 905 nm) and its efficacy in the treatment of chronic nonspecific low back pain is still unknown.

This work aims to study the effects of MSL laser therapy on pain, disability disability, lumbar ROM and muscle activity in a homogeneous group of patients with from chronic nonspecific low back pain. Although the literature shows that the combination of exercise with laser therapy yields better results in terms of both pain reduction and functional recovery, in this study we chose not to use any combination of treatments, in order to evaluate the effectiveness of MLS laser therapy alone in the treatment of chronic nonspecific low back pain.

To isolate the specific results of MLS laser therapy, it is intended to compare it with a placebo, represented by a device apparently identical in morphology and behavior to that delivering the laser and emitting visible light of similar appearance, by means of a clinical trial double-blind prospective randomized controlled trial. The double-blind design is adhered to because the type of laser therapy employed with the protocol followed, despite the effects tissue biology highlighted in the literature, is not able to make the patient feel any heat sensation during the session. 31 This is the first study in the literature aimed at analyzing the possible effects determined by the use of MLS laser therapy in chronic nonspecific low back pain: this investigation is conducted with an integrated methodology, using standardized and validated measures for pain intensity and disability, combined with kinematic and electromyography of high technological value.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (> 3 months)
* Lack of effectivness of previous conservative therapies for low back pain
* Body mass index < 30
* Preserved cognitive ability to fully understand and observe indications received by medical personnel
* Ability to understand and give an informed consent

Exclusion Criteria:

* Spine surgery
* Spinal hernia
* spondylolisthesis
* Spinal infections
* Severe spine deformities
* Neural diseases
* Rheumatic diseases
* Diabetes
* Psychiatric diseases
* Vascular diseases
* Cancer
* Infectious diseases
* Kidney stones
* Skin abrasion
* Pregnancy or breastfeeding
* Recent injuries
* Known sensibility to Laser therapy
* Epilepsy
* Anticoagulant therapy
* Pacemaker
* hemorrhagic diathesis
* Photosensitizing drugs
* Kown Photosensibility
* Low back Tattoos
* Steroid injections in the previous 3 weeks
* Antinflammatory or pain drugs
* HIV positive
* Neuro-stimulation implanted systems
* Tissue with ischemia in the low back

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Low back pain | At baseline (T0)
  VAS, Visual Analogic Scale minimum 0 (the best) and maximum 10 (the worst)
Low back pain | 3 weeks (T1)
  VAS, Visual Analogic Scale minimum 0 (the best) and maximum 10 (the worst)
Low back pain | One month by the end of the intervention (T2)
  VAS, Visual Analogic Scale minimum 0 (the best) and maximum 10 (the worst)

SECONDARY OUTCOMES:
Disability | At baseline (T0)
  Roland-Morris questionnaire
Disability | 3 weeks (T1)
  Roland-Morris questionnaire
Disability | One month by the end of the intervention (T2)
  Roland-Morris questionnaire
Pain and Disability | At baseline (T0)
  Oswestry disability questionnaire
Pain and Disability | 3 weeks (T1)
  Oswestry disability questionnaire
Pain and Disability | One month by the end of the intervention (T2)
  Oswestry disability questionnaire

OTHER OUTCOMES:
Trunk kinematics | At baseline (T0)
  Degree of trunk flexion and velocity of the flexion measured with an accelerometer
Trunk kinematics | 3 weeks (T1)
  Degree of trunk flexion and velocity of the flexion measured with an accelerometer
Trunk kinematics | One month by the end of the intervention (T2)
  Degree of trunk flexion and velocity of the flexion measured with an accelerometer
Low back muscles activation | At baseline (T0)
  Flexion-relaxation phenomenon assessed by means of surface EMG electrodes placed over the longissimus dorsi and the multifidus muscles
Low back muscles activation | 3 weeks (T1)
  Flexion-relaxation phenomenon assessed by means of surface EMG electrodes placed over the longissimus dorsi and the multifidus muscles
Low back muscles activation | One month by the end of the intervention (T2)
  Flexion-relaxation phenomenon assessed by means of surface EMG electrodes placed over the longissimus dorsi and the multifidus muscles

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Benedetti, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS-Istituto Ortopedico Rizzoli, Bologna, Italy